CLINICAL TRIAL: NCT00183482
Title: Family Cognitive Behavioral Prevention of Depression in Children of Parents With a History of Major Depressive Disorder
Brief Title: Family Cognitive Behavioral Therapy for Preventing Depression in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Bruce Compas, Patricia and Rodes Hart Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH100258 (NIH); R01MH100258 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Depression
Keywords: Parents; Child; Stress; CBT
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Repeated measures ANCOVA design.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcome assessors are masked to condition of participants.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Group Cognitive Behavioral (Experimental): The intervention is a family group cognitive behavioral program for families of parents with a history of depression to teach parenting skills to parents and coping skills to children.
  Interventions: Behavioral: Family Group Cognitive Behavioral
- Written Information (Active Comparator): The comparison arm involves providing written information about depression and stress to parents with a history of depression and their children.
  Interventions: Behavioral: Written Information

INTERVENTIONS:
Behavioral: Family Group Cognitive Behavioral — Groups of families receive training in parenting and children learn about coping in ten weekly sessions and then three monthly sessions
  Arms: Family Group Cognitive Behavioral
Behavioral: Written Information — Families are mailed written materials that describe depression and stress in families with a depressed parent.
  Arms: Written Information

SUMMARY:
This study will determine the effectiveness of cognitive behavioral therapy (CBT) versus educational treatment in preventing depression in the children of parents with a history of depression.

DETAILED DESCRIPTION:
Depression is a serious condition that can affect a person's work, relationships, and quality of life. Studies have shown that children of depressed parents are at a higher risk for developing depression than those whose parents have not experienced depression. Safe and effective treatments that can help prevent children of depressed parents from becoming depressed are needed. This study will compare CBT to depression education to determine which is more effective in preventing depression in the children of depressed parents.

Families will be randomly assigned to receive weekly sessions of either CBT or depression education for 12 weeks. Parents in the CBT group will be taught skills to more effectively raise their children and to better manage their depressive symptoms; their children will be taught skills to cope with the stress of their parents' depression. Families in the education group will be informed about the ways that depression can affect individuals with depression and their families.

Study visits will occur at study entry and at Week 12. Several follow-up visits will occur for up to 2 years after the interventional part of the study. At each visit, a clinician will make direct observations of the depressed parent's interaction with his or her children. In addition, families will be interviewed and will complete questionnaires about the parent's depressive symptoms and family interaction.

ELIGIBILITY:
Inclusion Criteria for Participating Families:

* Families with at least one parent with a history of depression during the life of his or her child
* Families with at least one child between the age of 10 and 15
* Parent or guardian willing to provide informed consent for participating children

Exclusion Criteria for All Participants:

* Parent with bipolar disorder or schizophrenia
* Child with conduct disorder or pervasive developmental disorder

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Internalizing and Externalizing symptoms in children | 12 months
  Child Behavior Checklist; Youth Self-Report; Internalizing and Externalizing Problems; Minimum T score = 40; Maximum T score = 80; Higher scores reflect worse outcome

SECONDARY OUTCOMES:
Depressive symptoms in parents | 12 months
  Patient Health Questionnaire - 9; Total Depression Symptoms; Minimum score = 0; Maximum score = 27; Higher scores reflect worse outcomes
Coping skills of children | 12 months
  Responses to Stress Questionnaire; Secondary control coping scale; Minimum score = 4; Maximum score = 16; Higher scores reflect better outcomes
Parenting skills of parents | 12 months
  Parent-child interaction coded
Onset of depressive disorders in children | 12 months
  Interviews

CONTACTS AND LOCATIONS:
Overall Officials: Bruce E. Compas, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Ciriegio AE, Pine AE, Cole DA, McKee LG, Forehand R, Compas BE. Mediators of a randomized controlled trial of a preventive intervention for youth of parents with depressive disorders. J Consult Clin Psychol. 2025 Jan;93(1):1-13. doi: 10.1037/ccp0000928. PMID 39786802